CLINICAL TRIAL: NCT06885710
Title: Safety and Efficacy of Hepatitis B Virus (HBV)-Specific T Cell Receptor (TCR)-T Cell Therapy Combined With Nucleos(t)Ide Analogues (NAs) in HBeAg-Positive Chronic Hepatitis B Patients
Brief Title: HBV-Specific TCR-T Cell Therapy Combined With Nucleos(t)Ide Analogues in Chronic Hepatitis B Patients
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: Guangzhou Lion TCR Co Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTCR-CHB-1-1
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Chronic Hepatitis b
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- LioCyx-M (Autologous T-cells transfected with mRNA encoding HBV antigen specific TCR) (Experimental): Escalating doses of LioCyx-M from 5×10E05 to 50×10E06 cells/kg body weight (BW), administered every two weeks.
  Interventions: Biological: LioCyx-M

INTERVENTIONS:
Biological: LioCyx-M — Each patient will receive LioCyx-M infusion every one or two weeks, while continuing their existing nucleos(t)ide analog treatment.

SUMMARY:
This is a open-label study to evaluate the safety and efficacy of autologous T-cells transfected with messenger ribonucleic acid (mRNA) encoding Hepatitis-B virus (HBV) antigen specific T cell receptor (TCR) in combination with nucleos(t)ide analogues (NAs) in HBeAg-positive and negative chronic hepatitis B patients.

ELIGIBILITY:
Inclusion Criteria:

* CHB infection (Serum HBsAg-positive for ≥ 6 months)
* Serum HBeAg-positive or negative
* HLA class 1 profile matching HLA-class I restriction element of the available T cell receptors (restricted by either HLA-A*02:01, A*11:01 or A*24:02).
* Liver biopsy, Fibroscan or equivalent test obtained within the past 6 months demonstrating liver disease consistent with chronic HBV infection without evidence of bridging fibrosis or cirrhosis (≥Metavir 3).

Exclusion Criteria:

* History or other evidence of chronic liver disease unrelated to HBV infection (e.g., hemochromatosis, autoimmune hepatitis, alcoholic liver disease, toxin exposure, thalassemia, non-alcoholic fatty liver disease)
* Decompensated liver function, such as Child-Pugh grade B or C, or clinical signs of decompensated liver function like ascites and varices
* Positive HIV test result
* History or suspected diagnosis of hepatocellular carcinoma, or AFP at screening > 20 ng/mL (if AFP > 20 ng/mL, a liver scan result is required to exclude hepatocellular carcinoma)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2024-12-31 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Assessments of adverse events | Start of treatment until 28 days post last dose
  To evaluate the safety of LioCyx-M

SECONDARY OUTCOMES:
Changes in HBeAg levels | Up to 1 year after last dose
  To evaluate the anti-viral efficacy of LioCyx-M
Changes in HBeAb levels | Up to 1 year after last dose
  To evaluate the anti-viral efficacy of LioCyx-M
Changes in HBsAg levels | Up to 1 year after last dose
  To evaluate the anti-viral efficacy of LioCyx-M

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, China